CLINICAL TRIAL: NCT05780905
Title: Effects of Semaglutide on Intracranial Blood Flow and Brain-Barrier Permeability in Type-2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Francis Kim, Professor, Division of Cardiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: STUDY00016594; U1111-1271-3352 (Other Grant/Funding Number: Novo Nordisk US)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Stroke (CVA) or Transient Ischemic Attack
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Stroke; Ischemic Attack, Transient | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind and placebo controlled MRI study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to placebo for 1 year.
  Interventions: Other: Placebo
- Active (Active Comparator): Subjects randomized to semaglutide for 1 year.
  Interventions: Drug: Semaglutide Auto-Injector

INTERVENTIONS:
Drug: Semaglutide Auto-Injector — Subjects have an equal chance of receiving semaglutide or placebo. Which treatment subjects receive is decided at random by a computer (purely by chance, like the tossing of a coin). Neither subjects, Study Site personnel nor image reviewers will know which treatment subjects are assigned to. The study drug must be taken weekly. The subject's other medications may be changed by the study's un-blinded Endocrinologist.
  At baseline subject will receive and take home 0.25mg injector for use 3 more times. They will be given a 0.5mg injector and a 1mg injector for use beginning 5 and 9 weeks from baseline respectively.
  The target dose for subjects is 1mg per week up to the 52 week treatment duration.
  Other Names: ozempic
  Arms: Active
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A human subjects research study, the primary purpose of which is to assess the EFFECTS OF SEMAGLUTIDE ON INTRACRANIAL BLOOD FLOW AND BLOOD-BRAIN BARRIER PERMEABILITY IN TYPE-2 DIABETES (T2D) through testing of the intervention on patients in a clinical setting. The study will randomize subjects with diabetes to either semaglutide or matching placebo. Magnetic resonance images will be primary endpoint measured at baseline and at one year to assess effect of this FDA approved medication.

Given the available evidence supporting the neuroprotective effect of this drug class and stroke reduction with semaglutide, and the investigators preliminary data showing that T2D had significantly reduced total number of distal arterial branches in the brain than non-T2D, the investigators expect treatment with semaglutide will be associated with improved intracranial blood flow condition.

DETAILED DESCRIPTION:
The investigators preliminary data showed that T2D had significantly reduced total number of distal branches as assessed using the investigators quantitative magnetic resonance angiography (MRA) feature measurement method (iCafe) than non-T2D. This reduction represents a decrease in intracranial blood flow condition and can be an indication for ischemia. Clinical trial showed that semaglutide reduces stroke incidence in T2D. The investigators are conducting a randomized, double blind and placebo-controlled study to investigate the biological basis of the observed stroke reduction with semaglutide by demonstrating semaglutide can improve intracranial blood flow condition and reduce bloodbrain barrier (BBB) permeability. The investigators working hypothesis is that it is known that semaglutide has beneficial effects on T2D, therefore, it improves endothelial function for a better cerebral flow condition. However, semaglutide may also improve cerebral flow independently from glucose lowering. Together, the improved cerebral flow condition results in stroke reduction. In order to investigate the independent effects of semaglutide on intracranial blood flow condition and BBB permeability, the investigators will have a designated diabetes care specialist unblinded to the study randomization to carry out glucose management to achieve HbA1C<7.5% for both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 40-65 years of age
2. Subjects with type-2 diabetes >= 3 years and HbA1C 7%-10% with blood sugar control medications including insulin, metformin, sulfonylureas, or SGLT2 inhibitors
3. Medically stable
4. Has not received any investigational drug in the past 6 months
5. Willing to participate and sign informed consent.

Exclusion Criteria:

1. Contraindication to MRI or contrast agent
2. eGFR<45 mL/min/1.73m2 (eGFR is a measurement of kidney function)
3. Currently treated with glucagon-like peptide-1 receptor antagonist (same drug class as study intervention)
4. Unable to perform home-glucose monitoring
5. Currently need more than 100 units of insulin daily
6. Uncontrolled hypertension with systolic blood pressure (SBP)>180 mmHg or diastolic blood pressure (DBP)>100 mmHg
7. LDL-C>130 mg/dL or not on stable statin therapy in the past 6 months
8. Treatment with pioglitazone in the past 3 months
9. History of pancreatitis
10. History of myocardial infarction, stroke or transient ischemic attack
11. History or family history of Medullary Thyroid Carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
12. Hypersensitivity to semaglutide or any of the product components
13. Participating in other clinical trial
14. Women of child-bearing potential (ie, those who are not chemically or surgically sterilized or who are not post-menopausal) who have a positive pregnancy test at enrollment or who are breastfeeding or who plan to become pregnant in the next 15 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial blood flow (IBF) | Approximately 12 Months
  measured as total length and number of distal vessels
bloodbrain barrier Ktrans | Approximately 12 Months
  measured by dynamic contrast-enhanced MRI

SECONDARY OUTCOMES:
Inflammatory markers | Approximately 12 Months
  hsCRP, interleukin-6 and tumor necrosis factor -a

CONTACTS AND LOCATIONS:
Overall Officials: Francis Kim, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington - Harborview Medical Center, Seattle, Washington, United States